CLINICAL TRIAL: NCT07327866
Title: Incidence of Post-Spinal Anaesthesia Hypotension in Caesarean Delivery: A Randomized Trial of Classic Versus Sequential Spinal Technique
Brief Title: Comparison of Classic and Sequential Spinal Techniques for Preventing Hypotension During Cesarean Delivery.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC. 16.10.2025
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Caesarean Delivery; Hypotension Postprocedural
Keywords: Classic; Sequential Spinal Technique

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic group (Experimental): In the classic group, patients will receive a total intrathecal dose of 12.5 mg hyperbaric bupivacaine 0.5% (2.5 mL) combined with fentanyl 20 µg, administered as a single injection. Immediately after completion of the injection, the patient will be positioned supine with a 15° left lateral tilt to minimize aortocaval compression and facilitate uniform spread of the anesthetic solution.
  Interventions: Procedure: Classic group
- Sequential group (Active Comparator): In the sequential (fractionated) group, patients will receive the intrathecal dose in two fractions. While in the sitting position, the first fraction consisting of 7.5 mg (1.5 mL) of hyperbaric bupivacaine 0.5% combined with fentanyl 15 µg will be administered. After waiting for 60 seconds, the remaining 5 mg (1 mL) of hyperbaric bupivacaine and an additional 5 µg of fentanyl will be injected, either through the same intrathecal needle (if kept in place) or following careful reinsertion according to institutional practice. Immediately after completing the injection, the patient will be positioned supine with a 15° left lateral tilt to optimize maternal hemodynamics and ensure even distribution of the anesthetic solution.
  Interventions: Procedure: Sequential group

INTERVENTIONS:
Procedure: Classic group — In the classic group, patients will receive a total intrathecal dose of 12.5 mg hyperbaric bupivacaine 0.5% (2.5 mL) combined with fentanyl 20 µg, administered as a single injection. Immediately after completion of the injection, the patient will be positioned supine with a 15° left lateral tilt to minimize aortocaval compression and facilitate uniform spread of the anesthetic solution.
  Arms: Classic group
Procedure: Sequential group — In the sequential (fractionated) group, patients will receive the intrathecal dose in two fractions. While in the sitting position, the first fraction consisting of 7.5 mg (1.5 mL) of hyperbaric bupivacaine 0.5% combined with fentanyl 15 µg will be administered. After waiting for 60 seconds, the remaining 5 mg (1 mL) of hyperbaric bupivacaine and an additional 5 µg of fentanyl will be injected, either through the same intrathecal needle (if kept in place) or following careful reinsertion according to institutional practice. Immediately after completing the injection, the patient will be positioned supine with a 15° left lateral tilt to optimize maternal hemodynamics and ensure even distribution of the anesthetic solution.
  Arms: Sequential group

SUMMARY:
Given the clinical importance of maternal hypotension, the potential advantages of sequential spinal dosing warrant formal evaluation in a prospective, adequately powered randomized controlled trial. We therefore designed this study to compare the incidence of post-spinal hypotension between the classic single-shot spinal and the sequential fractionated spinal techniques in elective cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Adult women aged 18-45 years.
* ASA physical status II-III.
* Scheduled for elective cesarean section under standardized spinal anesthesia.

Exclusion Criteria:

* Allergy to local anesthetics.
* Emergency cesarean section.
* Contraindication to spinal anesthesia (e.g., coagulopathy, infection at the puncture site).
* Preexisting hypertension on medication or pre-eclampsia with severe features.
* Known cardiac disease accompanied by hemodynamic instability.
* Allergy to study drugs.
* Fetal distress or non-reassuring cardiotocography (CTG).
* BMI >40 kg/m².
* Refusal to sign informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Caesarean Delivery
Enrollment: 94 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-spinal hypotension | Assessed during the first 15 minutes after the intrathecal injection.
  Occurrence of maternal hypotension within 15 minutes after intrathecal injection, defined as a systolic blood pressure (SBP) decrease greater than 20% from baseline or an absolute SBP below 90 mmHg. This outcome directly measures the hemodynamic stability achieved by each spinal technique.

SECONDARY OUTCOMES:
Time to first hypotensive episode | Measured continuously for 15 minutes following the intrathecal injection.
  The interval between the time of intrathecal injection and the first recorded episode of hypotension. This reflects how long each technique maintains stable blood pressure before any drop occurs.
Number of hypotensive episodes | Assessed within 15 minutes after intrathecal injection.
  The total count of discrete hypotensive events occurring within the observation period after spinal anesthesia. This indicates the frequency and severity of blood pressure fluctuations.
Total vasopressor dose | Assessed within 15 minutes after spinal administration.
  The total amount of phenylephrine and/or ephedrine administered to correct hypotension during the observation period, serving as an indirect measure of hemodynamic stability.
Maximal sensory block level and time to T4 | Evaluated from injection until block stabilization within 20 minutes.
  Determines the highest dermatomal sensory level achieved and the time required to reach the T4 level, indicating block quality and onset characteristics of the anesthetic technique. Maximal sensory block level is assessed by testing loss of sensation to cold or pinprick over the trunk in a cephalad-caudal direction and mapping the highest blocked dermatome (e.g., using an alcohol swab or pin along the midline and comparing to known dermatomal levels such as T4 at the nipple line). Time to T4 is measured as the interval in minutes from completion of intrathecal injection to the first assessment at which loss of sensation reaches the T4 dermatome, documented with the same stimulus and dermatomal map.
Maternal nausea and vomiting | Monitored intraoperatively up to delivery.
  Incidence of intraoperative nausea or vomiting related to hypotension or anesthetic effect.
Maternal satisfaction | Assessed after delivery before discharge from recovery.
  Maternal satisfaction will be evaluated using a 5-point Likert scale addressing analgesia adequacy, comfort, and overall anesthesia experience. Each participant will rate her satisfaction as follows: 1 for "very dissatisfied," indicating poor pain control and significant discomfort; 2 for "dissatisfied," reflecting partial relief with ongoing discomfort; 3 for "neutral," denoting acceptable but unremarkable pain relief; 4 for "satisfied," representing good pain control with minimal discomfort; and 5 for "very satisfied," indicating excellent analgesia and a fully positive anesthesia experience.
Neonatal outcomes (Apgar scores and umbilical artery pH) | Determined immediately after delivery (Apgar at 1 and 5 minutes; pH from cord sample at birth).
  Measures neonatal wellbeing through 1-minute and 5-minute Apgar scores and umbilical artery blood pH to assess the effect of maternal hemodynamics on fetal oxygenation.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared upon a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP